CLINICAL TRIAL: NCT03260712
Title: Open-label First Line, Single-arm Phase II Study of CisGem Combined With Pembrolizumab in Patients With Advanced or Metastatic Biliary Tract Cancer
Brief Title: Pembrolizumab in Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1607-GITCG / ABC-09
Record Dates: First submitted 2017-08-08; First posted 2017-08-24 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Biliary Tract Cancer; Metastatic Cancer; Advanced Cancer; Gallbladder Cancer
Keywords: biliary tract cancer; metastitic cancer; advanced cancer; pembrolizumab; cisplatin; gemcitabine; gallbladder cancer
MeSH Terms: conditions — Biliary Tract Neoplasms; Neoplasm Metastasis; Gallbladder Neoplasms | interventions — pembrolizumab; spartalizumab; Cisplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- CisGem + pembrolizumab (Experimental): Patients will be enrolled in the experimental arm and will receive CisGem [25mg/m2 cisplatin + 1000mg/m2 gemcitabine, on days 1 and 8 of a 21 day cycle] plus 200 mg pembrolizumab (fixed dose) on day 1 of a 21 day cycle.
  Interventions: Drug: Pembrolizumab; Drug: Cisplatin; Drug: Gemcitabine

INTERVENTIONS:
Drug: Pembrolizumab — The dose of pembrolizumab in this trial is 200 mg Q3W.
  Other Names: Anti-PD-1
Drug: Cisplatin — 25mg/m2 cisplatin on days 1 and 8 of a 21 day cycle
Drug: Gemcitabine — 1000mg/m2 gemcitabine on days 1 and 8 of a 21 day cycle

SUMMARY:
This is a single-arm, multi-centre, phase II study in biliary tract cancer (BTC) patients. The main objective is to detect an increase in progression-free survival rate at 6 months (according to RECIST version 1.1) from 60% in patients with BTC treated with standard chemotherapy (CT) approach to 75% when treated with CT combined with pembrolizumab.

DETAILED DESCRIPTION:
Primary endpoint: PFS rate at 6 months according to RECIST 1.1.

Secondary endpoints:

* Best overall response rate (according to RECIST 1.1 and iRECIST)
* Response duration and stable disease duration (according to RECIST 1.1 and iRECIST)
* PFS rate at 6 months according to iRECIST
* PFS according to RECIST 1.1 and iRECIST
* Overall survival (OS)
* Toxicity of treatment (Common Toxicity Criteria CTCAE 5.0)
* Safety analysis: A safety analysis will be done when at least 10 patients have completed at least one cycle of the three- drug combination.

Events of clinical interest for this safety analysis are the following:

* At least Grade 2 or higher CTCAE 5.0 signs of acute renal failure
* Grade 3 or 4 liver dysfunction defined as elevation of liver transaminases (AST and ALT) and alkaline phosphatase, increased bilirubin
* Grade 3 or 4 gastrointestinal disorders specifically colitis, diarrhea and stomatitis
* Grade 3 or 4 dyspnea, dry cough and pneumonia
* Grade 3 or 4 sepsis
* Grade 3 or 4 skin toxicity If 4 out of these 10 patients experience any of the above, this will trigger an IDMC review. This cut-off is based on: 1) previous ABC-02 study where 57% of patients experienced a grade 3 or 4 toxicity at 12 weeks of treatment; and 2) KEYNOTE 028 where 17% of patients experienced grade 3 or 4 toxicity The primary analysis of efficacy endpoints will be performed in the protocol population.
* PFS rate at 6 months will be estimated using Kaplan Meier estimate at the time point of interest. The lower bound of the one-sided 90% confidence interval (CI) will be calculated by Greenwood's estimation of the standard deviation. If the lower bound of the one-sided 90% CI is above 60%, it will be concluded that the new treatment is effective enough to warrant further evaluation in a phase III trial. Assuming exponential distributions for both PFS and for the risk of drop-out, power with a total sample size of 50 patients when the primary test is performed using Kaplan Meier analyses will be around 82% for a drop-out rate of 5% at 6 months and still above 80% for a drop-out rate of 10% at 6 months. The one-sided type I error will be respectively 9.33% and 9.02%.
* PFS rate at 6 months according to iRECIST will be estimated using Kaplan Meier estimate and the one-sided 90% confidence interval (CI) will be calculated by Greenwood's estimation of the standard deviation.
* BOR rate according to RECIST 1.1 and iBOR rate according to iRECIST will be displayed (point estimate) with their exact two-sided 95% confidence intervals. Response duration and stable disease duration according to RECIST 1.1 and iRECIST will be graphically displayed using swimmer plots and bar charts.
* Progression free survival according to RECIST 1.1 and iRECIST and overall survival curves will be estimated using the Kaplan-Meier technique. The safety analyses will be performed in the Safety population. The worst toxicity grade per patient over the treatment period according to the CTCAE criteria version 5.0 will be displayed.

ELIGIBILITY:
Inclusion Criteria:

* A histopathological / cytological diagnosis of non-resectable or recurrent / metastatic biliary tract carcinoma (intra- or extra-hepatic) or gallbladder
* Availability of archival FFPE tumor tissue for biobanking
* Measurable disease by CT/MRI (RECIST 1.1) within 28 days of enrollment
* ECOG performance status 0, 1
* Age ≥ 18 with estimated life expectancy >3 months
* Adequate hematological function: screening labs should be performed within 14 days (± 3 days) prior to enrollment:
* Hemoglobin ≥ 10 g/dl* (prior transfusions for patients with low hemoglobin are allowed)
* White blood cell (WBC) ≥ 3.0 x 109/L
* Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Platelet count ≥ 100 x 109/L
* Adequate liver function: screening labs should be performed within 14 days (± 3 days) prior to enrollment:
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN)
* ALT and/or AST & alkaline phosphatase ≤ 5 x ULN
* Adequate renal function: screening labs should be performed within 14 days (± 3 days) prior to enrollment:
* Serum creatinine < 1.5 x ULN
* and a calculated GFR ≥ 45 mL/min (using Cockcroft-Gault formula). If the calculated GFR is below 45 mL/min, isotope EDTA confirmation of adequate renal function is required (see Appendix F). If isotope EDTA methods are not available, then a 24-hour urine creatinine clearance can be used.
* Adequate coagulation: screening labs should be performed within 14 days (± 3 days) prior to enrollment:
* International Normalized Ratio (INR) or Prothrombin Time (PT): ≤ 1.5xULN unless patient is receiving anticoagulant therapy as long as PT or Partial Thromboplastin Time (PTT) is within therapeutic range of intended use of anticoagulants
* Adequate biliary drainage with C-reactive protein (CRP) levels in normal ranges (based on institution's standard): screening labs should be performed within 14 days (± 3 days) prior to enrollment
* Patient is not currently participating and receiving study therapy or has not participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks prior to enrollment
* Women of child bearing potential (WOCBP) must have a negative serum (or urine) pregnancy test within 72 hours prior to the first dose of study treatment.
* Patients of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the study treatment period and for at least 6 months after the last study treatment. A highly effective method of birth control is defined as those which result in low failure rate (i.e. less than 1% per year) when used consistently and correctly. Such methods include:
* Combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
* Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
* Intrauterine device (IUD)
* Intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion
* Vasectomised partner
* Sexual abstinence. Note: abstinence is acceptable if this is established and preferred contraception for the patient and is accepted as a local standard.
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 120 days after the last study treatment.
* Before patient enrollment, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Patients with ascites grade 2 or higher
* Child Pugh B or C hepatic impairment
* Incomplete recovery from previous surgery or unresolved biliary tract obstruction
* Active infection requiring therapy. Antibiotic treatment should have been completed 5 days before enrollment
* Patients who are candidates for curative surgery
* History of (non-infectious) pneumonitis that required steroids or current pneumonitis. No history of or current interstitial lung disease
* Active autoimmune disease that has required systemic treatment in past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Diagnosis of immunodeficiency, systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment
* Known history of human immunodeficiency virus (HIV), active Hepatitis B or Hepatitis C
* Patients with hyperthyroidism or hypothyroidism unless stable on hormone replacement
* History of another malignancy or a concurrent malignancy. Exceptions include patients who have been disease-free for 5 years, or patients with a history of completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible, for example cervical cancer in situ.
* Patients who received treatment with live vaccines within 30 days prior to the first dose of study medication. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, shingles, yellow fever, seasonal flu, H1N1 flu, rabies, BCG and typhoid vaccine.
* Prior treatment with any anti-CTLA4 monoclonal antibody or anti-PD-1, or PD-L1 or PD-L2 agent. Examples of PD-1 inhibitors (include, but are not limited to): pembrolizumab (Merck); Nivolumab (also known as BMS-936558, MDX-1106, ONO-4538) (Bristol-Myers Squibb); Pidilizumab (CT-11) (Cure-Tech/Teva); and AMP-224 (Amplimmune). Examples of PD-L1 inhibitors (include, but are not limited to): BMS-936559 (also known as MDX-1105) (Bristol-Myers Squibb); MPDL3280A (also known as RG7446) (Roche Genentech); and MEDI4736 (MedImmune).
* Prior systemic chemotherapy for locally advanced or metastatic disease.
* Prior adjuvant chemotherapy is allowed if the last treatment was completed at least 6 months before trial entry and neither gemcitabine nor cisplatin were given. Also the following treatment modalities are allowed within the rules described (provided there has been a full recovery):
* Surgery - patients may have undergone a non-curative operation (i.e. R2 resection [with macroscopic residual disease] or palliative bypass surgery only). Patients who have previously undergone curative surgery, must have evidence of non-resectable disease relapse requiring systemic chemotherapy prior to study entry.
* Radiotherapy - patients may have received prior radiotherapy (with or without radiosensitising low-dose chemotherapy) for localised disease. However, there must be clear evidence of disease progression prior to inclusion in this study.
* Photodynamic therapy (PDT) for localized disease only with no evidence of metastatic disease - patients may have received prior PDT, provided the patient has fully recovered and at least 28 days have elapsed since the PDT and there is clear evidence of disease progression at the local site or disease or at a new metastatic site.
* PDT for localised disease to relieve biliary obstruction in the presence of metastatic disease - patients may have received prior PDT provided the patient has fully recovered and at least 28 days have elapsed since the PDT. Patients may enter trial provided the non-PDT treated lesion(s) only are followed for response assessment.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before enrollment in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Detection of progression-free survival (PFS) rate at 6 months defined according to RECIST 1.1. | At 6 months
  The main objective is to detect an increase in progression-free survival (PFS) rate at 6 months (according to RECIST version 1.1) from 60% in patients with BTC treated with standard chemotherapy approach to 75% when treated with CT combined with pembrolizumab.

SECONDARY OUTCOMES:
Best overall response rate (according to RECIST 1.1) and overall response | Up to 120 days after last administration of Pembrolizumab
  Assessing both short term and long term outcome of patients receiving this combined treatment
Toxicity (according to CTCAE 4.03) | Up to 120 days after last administration of Pembrolizumab
  Establishing the safety of standard chemotherapy combined with pembrolizumab in these patients
Progression free survival rate at 6 months according to iRECIST | At 6 months

OTHER OUTCOMES:
Immunological response (cytokines, lymphocyte phenotype, immunoglobulins) | Up to 2 years after start of study treatment
  Assessment of immunological responses (cytokines, lymphocyte phenotype, immunoglobulins)
Pathological predictive factors for response and toxicity (TCR Sequencing, FACs, RNASeq, nanostring) | Up to 2 years after start of study treatment
  Evaluation of pathological predictive factors for response and toxicity
Clinical predictive factors for response and toxicity (TCR Sequencing, FACs, RNASeq, nanostring) | Up to 2 years after start of study treatment
  Evaluation of clinical predictive factors for response and toxicity
Biomarkers predictive of response and toxicity (protein profiling, HLA typing) | Up to 2 years after start of study treatment
  Evaluation of biomarkers for prediction of response and toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Markus Moehler, Prof. Dr., Study Chair — Johannes Gutenberg Universitaetskliniken - Mainz University Medical Center
Locations (7):
- Germany (2):
  - Universitaetsklinikum Leipzig UCCL-Krebszentrum, Leipzig
  - Universitaetsmedizin der Johannes Gutenberg Universitaet Mainz-University Medical Center, Mainz
- Spain (2):
  - Vall d'Hebron Institut Oncologia, Barcelona
  - Hospital Universitario 12 De Octubre, Madrid
- United Kingdom (3):
  - University College London Hospitals NHS Foundation Trust - University College Hospital, London
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham